CLINICAL TRIAL: NCT05256069
Title: Sex-related Differences in Sympathetic Vascular Transduction in the Setting of Hypoxemia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Jacqueline K Limberg, PhD, Assistant Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2087402
Record Dates: First submitted 2022-02-14; First posted 2022-02-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Vasodilation; Hypoxia
MeSH Terms: conditions — Aneurysm; Hypoxia | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypoxia Exposure (Experimental): Men and women will be exposed to isocapnic hypoxia. Participants will wear a mask and systemic oxygen levels will be titrated to attain hypoxemia as assessed by pulse oximetry.
  Interventions: Drug: Propranolol Pill; Drug: Placebo

INTERVENTIONS:
Drug: Propranolol Pill — Participants will receive a β-blockade (propranolol pill, 1 mg/kg dosed based on participant weight).
Drug: Placebo — Participants will receive a placebo in pill form.

SUMMARY:
The purpose of this project is to identify sex-related differences in the effect of hypoxia on sympathetic vascular transduction.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult men and women;
* 18-45 years of age;
* BMI 18-30 kg/m2;
* non-pregnant/non-breastfeeding;
* non-nicotine users;

Exclusion Criteria:

* Pregnancy, breastfeeding, hormonal contraceptives
* Diagnosed sleep apnea
* Current smoking/Nicotine use/drug use
* Nerve/neurologic disease
* Cardiovascular, hepatic, renal, respiratory disease
* Blood pressure ≥140/90 mmHg
* Diabetes, Polycystic ovarian syndrome
* Communication barriers
* Prescription medications
* Recent COVID-19 diagnosis with symptoms

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Forearm Blood Flow | Change from baseline to 5 minutes
  Measured with venous occlusion plethysmography (mL/dL/min)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline K Limberg, Ph.D., Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided